CLINICAL TRIAL: NCT04836624
Title: Co-designing Personalised Aids of Daily Living With Users With Chronic Conditions: a Feasibility Study
Brief Title: Co-designing Personalised Assistive Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Swansea Bay University Health Board (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RIO 008-21
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-05

CONDITIONS: Disability or Chronic Disease Leading to Disablement
Keywords: Co-design; Assistive technology; Assisitve Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Co-designing personalised aids of daily living (Experimental): Participants will be involved in up to 6 interactive sessions spread over 3 months with the researcher. Participants will work with the researcher to help develop their own assistive device to overcome challenges of daily living they experience.
  Interventions: Device: Co-designing of personalised aids of daily living

INTERVENTIONS:
Device: Co-designing of personalised aids of daily living — In the initial session the researcher will work with the participants to identify challenges in daily living for the device to overcome.
  In between sessions the researcher will design and manufacture different solutions which will then be sent out for the participant to trial. The participant will then meet with the researcher to and feedback on the device provided. Feedback from the user is used to alter and improve the design of the device; new device(s) are then , enabling the design to be adapted to the participants needs. The process of design changes and feedback forms an iterative loop. This is expected to continue for 4-5 appointments over a period of serveral months until a final design is agreed upon.
  After the device is issue, both qualitative and quantitative outcome measures are provided to participants to complete, including questionnaires and semi-structured interviews. .

SUMMARY:
Assistive technology is an important tool in helping people maintain independence, allowing them to actively participate in education, work, and society. If maximised to its full potential there would be significant health and wellbeing benefits for individuals, reduced reliance on formal health and social care services and reduced healthcare costs. However, current equipment is often unsuitable in meeting an individual's needs. Previous review work by the research team highlighted issues with the design, function, and service provision of assistive technology as barriers to its use. Two specific barriers, a lack of equipment customisation and a lack of end-user involvement in the provision process, are the focus of this work.

This research aims to assess a new method that provides personalised assistive technology to individuals. The method will actively engage participants to input into the design of their own assistive device(s) to help them overcome their challenges of daily living. This method will help enable the device to be customized to their needs, a process known as co-design. Participants will be recruited from Swansea Bay University Health Board with a range of long-term physical health conditions whose current needs are unable to be met by current standard and off-the-shelf assistive technology solutions. Participants must be aged 18+ and currently living within the community.

Participants will be involved in up to 6 interactive sessions spread over 3 months with the researcher. In the initial session the researcher will work with the participants to identify challenges in daily living for the device to overcome. In subsequent sessions, the researcher will design different solutions for the participant to try and feedback on, enabling the design to be adapted to the participants needs. Finally, the participants will evaluate the device provided through questionnaires and individual semi-structured interviews. This feedback will help assess the effectiveness of co-design and its feasibility to be incorporated into future NHS services.

DETAILED DESCRIPTION:
PROCEDURE:

1. Referral: Potential participants will be identified by a healthcare professional from their current care team and asked whether they would like to participate in the study. Potential participants will be provided with the participant information sheet and asked to consent if they would like their details to be referred onto the principal investigator.

   1.1 Arrange appointment: The principal investigator will telephone the potential participant to arrange an appointment to discuss their involvement in the research and gain consent. The consent form will be sent out to the participant (email or posted, depending on preference of participant).
2. Consent and eligibility [Virtual appointment]: The principal investigator will go through the participant information sheet with the participant and answer any questions they have about the study. The researcher will check they are eligible to take part in the study. If the participant is happy to be involved, they will be asked to sign the consent form and return it back to the researcher (either by email or posting back).
3. Initial assessment [Virtual appointment]: Through discussion with the participant, the researcher will gather relevant information to help identify their assistive technology needs. This will include information about their medical history and social context, likes and dislikes, current and any previous solutions used and challenges they faces in daily living. For each challenge identified, participants will be asked to score 1-5 about how important the challenge is to them and how difficult it is. This is for the Individually Prioritised Problem Assessment (IPPA) base-line measure. The researcher will complete the Client Service Receipt Inventory base-line measure with the participant to capture demographic information, information on heathcare services accessed in the previous 3 months and medication being taken.
4. Follow-up appointments, approximately 3-5 [Predominantly virtually, with face-to-face only if required]: In subsequent appointments the participant will meet with the researcher to discuss design ideas, provide feedback and agree on design changes for the devices(s) provided by the researcher to the participant. The participant will be asked to describe what they like/dislike about the current design and what changes they would make. The researcher may show design prototypes over video call to demonstrate how a device will work and to help facilitate gathering feedback.

   Following the appointment, the researcher will make design alterations, manufacture designs and post prototypes out for the participant to try. Appointments will be 2-3 weeks apart.
5. Device issue: Once the design has been refined to a level the participant and researcher are happy with, a final solution will be manufactured. The device will be sent out to the participant and the researcher will meet virtually with the participant to provide any necessary training and instructions for safe usage of the device.
6. Outcome measures [Virtually, same appointment as above]: The researcher will explain and go through the three different questionnaires being used as outcome measures for the study. The participant will be asked to score 1-5 the difficulty they now find the previously identified challenges (from initial assessment). For the two other measures, QUEST and PIADS [explained below], the researcher will either email or post out the questionnaires to the participant, preference of participant. Participants will be asked to complete and send back (email/post) once completed. Participants will be invited to complete the first of the semi-structured interviews with the researcher to obtain feedback on the co-design process and the device provided. Prior to beginning the interview, participants will be reminded it will be audio-recorded. If required, an additional appointment can be arranged to help the participant complete the questionnaires.
7. Three month follow-up feedback [Virtual appointment]: Participants will be invited to again complete and return the two questionnaires, QUEST and PIADS, to the researcher. Participants will complete the follow-up CSRI with the researcher. Participants will also be invited to undertake the second semi-structured interview to obtain feedback on the long-term use of device provided. Prior to beginning the interview, participants will be reminded it will be audio recorded Upon completion of the interview the participants involvement in the study will finish. Participants will be advised to contact the Rehabilitation Engineering Unit with any issues with their devices or further queriers about the research.

SETTING:

Due to COVID-19 pandemic, where possible the majority of appointments with occur virtually using a video consultation programme called Attend Anywhere. This will include assessing eligibility and gaining consent, initial assessment, follow-up appointments and the semi-structured interviews. Information on how to access an appointment through this will be provided to participants when they are invited to their first appointment.

Between appointments, the researcher will contact participants using telephone or email to arrange subsequent appointments. During the study, any devices for the participant to trial will be posted out to them. Training and/or instructions will be provided on how to use the device prior to it being sent out.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a long-term chronic condition
* Living in the community
* Age eighteen years or older
* Ability to actively engage in a co-design process, as determined by the referring clinician, including:
* Sufficient comprehension of language to engage in meaningful verbal dialogue with the researcher.
* Sufficient insight into their condition such that they understand their needs.
* Sufficient ability to communicate their needs.
* Sufficient ability to retain information between sessions
* Currently under the care of healthcare services within Swansea Bay University Health Board
* At least three-month post injury/diagnosis at the point of recruitment allowing time for spontaneous recovery and for the person to become aware of their difficulties and the implications of this on their lives

Exclusion Criteria:

* Receptive or expressive language difficulties, or extremely low memory function that may preclude people from engaging meaningfully
* Medically unstable, severe mental health or cognitive difficulties which may preclude meaningful engagement in the study.
* Not able to provide informed consent.
* Have insufficient access to the internet to engage virtually with the researcher through video conferencing software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Qualitative Feedback - Semi-structured interviews | At initial device issue and at 3-months post device issue
  Semi-structured questions will be used in individual interviews to facilitate an understanding of:
  * Any change the device(s) provided have had on the participants life
  * Identify components of the co-design methodology that participants like and dislike and changes to it in the future.
  * If co-design has changed any of the barriers to accessing and using assistive technology

SECONDARY OUTCOMES:
Quebec User Evaluation of Satisfaction with Technical Aids (QUEST 2.0) | At initial device issue and repeated at 3-months post device issue
  A 12-item outcome measure that assesses the user's satisfaction with both the device and service provided in supplying the device. For each item of the questionnaire, a 5-point scale is used, 1 being not satisfied at all and 5 being very satisfied.
Psychosocial Impact of Assistive Devices Scale (PIADS) | At initial device issue and repeated at 3-months post device issue
  A 26-item self-reported questionnaire to assess the effects of an assistive device on three sub-scales: competence, adaptability and self-esteem. For each item of the questionnaire, a 7-point scale is used, ranging from -3 (maximum negative impact) to 3 (maximum positive impact)
Individually Prioritised Problem Assessment (IPPA) | At initial appointment and repeated at initial device issue
  An instrument to assess the effectiveness of assistive technology provision in relation to activities the individual considers most relevant. The participant can select up to 7 problems they experience in everyday life. For each problem the participant assigns two scores, one for the importance of the activity and the second for the difficulty. Both scores are assigned using a 5 point scale: 1 not important to 5 most important and 1 not difficult to 5 too difficult to perform.
Client Service Receipt Inventory (CSRI) | Completed at the initial assessment and again at the 3-month follow-up assessment
  A tool used to capture and record information on health and social care services and resources used by study participants to help estimate the costs of services received. It will be used to calculate the economic cost changes associated with participation in the study.
  The inventory asks participants to idenfify the healthcare services they have accessed in the previous 3 months and any medication they are taking relevant to the health condition and challenges of daily living identified. It will also capture demographic information about the participants. The CRSI will measure any changes to services accessed, medication taken and demographic information as a result of participating in this study.

OTHER OUTCOMES:
Resources used | Through study completion, an average of 8 months.
  For each participant an estimate of the resources used and costs involved will be calculated. Costs will be calculated based on the number of person-hours required to engage participant and produce device, manufacturing time and material cost of all components required to produce the final device. This will include time for each appointment with the participant, time spent developing and changing the design, and time to create documentation required to comply with quality management system.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howard, PhD Student, Principal Investigator — Swansea University
Locations (1):
- Swansea Bay University Health Board, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No